CLINICAL TRIAL: NCT07257965
Title: A Clinical Study to Assess the Minimum Number of Infective Mosquito Bites to Achieve Malaria Infection in Healthy Thai Adults Using Controlled Human Plasmodium Vivax Infected Mosquito Challenge
Brief Title: Clinical Study to Assess Minimum Mosquito Bites for P. Vivax Infection in Thai Adults
Acronym: MIST4
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: MAL25001
Record Dates: First submitted 2025-11-14; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Plasmodium Vivax Infection
Keywords: Malaria; Mosquito bite; Plasmodium Vivax Infection
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Intervention Model Description: Three groups assigned sequencially. This is a single-centre, adaptive-design, Plasmodium vivax sporozoite-stage mosquito-bite Controlled Human Malaria Infection (CHMI) trial conducted in healthy, malaria-naïve Thai adults
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Number of mosquito bite (1 or 2 or 3) (Experimental): Number of mosquito bites assigned sequentially based on the adaptive design
  Interventions: Other: Mosquito bite (1 or 2 or 3)

INTERVENTIONS:
Other: Mosquito bite (1 or 2 or 3) — Successful feeding of 1, 2, or 3 Plasmodium vivax-infected mosquitoes

SUMMARY:
This study is a human challenge study to assess the minimum infective mosquito bite dose in a controlled human malaria Infection (via P. vivax sporozites) in healthy volunteers. The results will inform the development of a P. vivax mosquito-delivered CHMI trial platform, supporting safer and more accurate vaccine efficacy assessments. Conducting the trial in individuals genetically and immunologically similar to the target population will also enhance the relevance of findings to real-world endemic settings.

This study is funded by the UK Wellcome Trust. The grant reference number are Oxford/MORU: 212336/Z/18/Z and 212336/Z/18/A, and Mahidol University: 212336/A/18/Z and 212336/A/18/A.

DETAILED DESCRIPTION:
Controlled Human Malaria Infection (CHMI) has become an essential approach in the accelerated development of malaria vaccines and therapeutic interventions. This methodology involves the inoculation of human volunteers with malaria parasites, either via mosquito bites or direct administration of sporozoites or parasitized erythrocytes. CHMI facilitates the evaluation of vaccine and drug candidates in well-controlled early-phase clinical studies, enabling the selection of the most promising candidates for further evaluation in malaria-endemic regions.

While intravenous injections of parasites can be employed in such studies, the natural route of infection via mosquito bite has notable advantages, particularly in stimulating immune responses at the site of infection in the skin and closely mimic the natural infection process, allowing both liver and blood stage infections to develop. Additionally, mosquito-based challenge models provide a valuable platform for the evaluation of pre-erythrocytic (sporozoite) vaccine candidates. Effective sporozoite vaccines are expected to induce the production of serum antibodies capable of neutralizing sporozoites before they invade hepatocytes, thereby preventing liver-stage and blood-stage malaria.

Historically, numerous challenge studies using P. falciparum-infected mosquito bites or malaria parasite have been conducted in well-established research centers, including the Walter Reed Army Institute of Research, Sanaria Inc., the University of Maryland, Seattle Biomedical Research Institute, University of Oxford, and Radboud University Medical Centre. These studies have involved large cohorts, with over 45 trials involving P. falciparum-infected mosquitoes. However, studies utilizing P. vivax-infected mosquito bites have been fewer in number, with 8 trials conducted in regions such as Colombia, the UK, and Thailand.

P. vivax is the most prevalent malaria species outside of sub-Saharan Africa and represents a significant cause of malaria in countries such as Thailand. Given the substantial burden of P. vivax in Thailand and Southeast Asia, an international collaborative research team has proposed to advance the development and evaluation of P. vivax malaria vaccine candidates in an endemic region. This initiative is designed to include volunteers with genetic and immunological characteristics similar to those of the target population, thereby ensuring the relevance and applicability of the findings.

The first human challenge study in Thailand using P. vivax sporozoite infection known as "Malaria Infection Study in Thailand 1 (MIST1)," is currently being conducted at the Faculty of Tropical Medicine, an institution internationally recognized for its expertise in malaria research. The study aims to assess the feasibility and safety of P. vivax sporozoite human challenge in the local population. It represents a critical milestone in supporting the development and evaluation of effective malaria vaccines in regions where P. vivax is endemic.

Majority of malaria sporozoite challenge studies (75%, 39 out of 52 studies) have traditionally relied upon the bites of five infected mosquitoes to induce malaria. The rationale for using 5 mosquito bites is based on the extensive previous experience with P. falciparum, where sporozoite inoculated by fewer than five mosquitoes has led to inconsistent infections in malaria-naïve volunteers. However, this pattern does not appear to hold for P. Vivax-infected mosquito, as most studies demonstrated 100% infectivity rates using 2-4 mosquito bites and 5 mosquito bites. One study using P. Vivax-infected mosquito reported that 1 out of 18 participants did not develop malaria infection following a mosquito challenge. However, since antimalarial drug level were not measured in that study, the cause of this outcome remains inconclusive. Notably, no study used as few as one mosquito bite to induce P. Vivax malaria.

Individuals rarely bitten by more than one infected mosquito per night under natural condition, except in settings with very high malaria transmission intensity. In a very low transmission site on the Thai-Myanmar border a recent study reported a geometric mean of 57 sporozoites per mosquito (range 9-11,428). This compares to earlier studies in Africa and PNG where endemicity was higher and geometric means were >4000 (range 150-10,000). The probability of infection increases with the number of infectious bites. There are relatively little data on the number of sporozoites in naturally infected mosquitoes. It has been demonstrated that highly infected mosquitoes being more likely to have caused infection than lightly infected mosquitoes in a dose-response relationship.

The MIST1 study initially employed five mosquito bites to ensure consistent infection in a small cohort of six volunteers. However, using five mosquito bites may create an unrealistic challenge and could hinder the assessment of true vaccine efficacy. One out of five volunteers in the MIST1 study developed a relapsed Plasmodium vivax infection, suggesting that the standard challenge involving five Plasmodium vivax -infected mosquitoes might contribute to an overwhelming infection.

The primary aim of this study is to determine the minimum number of Plasmodium vivax-infected mosquito bites required to reliably induce malaria infection in healthy individuals. This study will begin with a challenge dose of two mosquito bites, as only a limited number of studies have evaluated challenge models using as few as 2-4 infected mosquitoes, and some involved small sample sizes. Furthermore, no study has used as few as one mosquito bite to induce P. vivax malaria.

The investigators aim to confirm whether 1 - 3 bites are sufficient to consistently induce P. vivax infection while maintaining a challenge model that more closely reflects natural transmission, avoids excessive parasite exposure, and could undermine the vaccine efficacy assessments. If at least one volunteer who receives two mosquito bites is not successfully infected, the investigators will increase the challenge dose to three bites. If at least one volunteer remains uninfected after three bites, the investigators will not escalate the challenge to four bites as reducing from standard five bites to four may not provide a meaningful advantage as suggested by the Steering Committee.

The study will provide important information for the development of P-vivax mosquito delivered CHMI trials platform, enabling a safer and more accurate assessment of vaccine efficacy in malaria research. Moreover, conducting this trial in a local population will enhance the applicability of the findings to rea-world endemic settings

ELIGIBILITY:
inclusion criteria

The volunteer must meet all of the following criteria to be eligible for the study:

1. Healthy adult aged 20 to 55 years with weight more than 50 kg.
2. No recent malaria infection.
3. Red blood cells positive for the Duffy antigen/chemokine receptor (DARC).
4. CYP2D6 alleles consistent with normal metaboliser status.
5. Normal level of Glucose-6-phosphate dehydrogenase (G6PD) enzyme activity by the WHO definition.
6. Women only: Must practice continuous effective contraception for the duration of study period until 3 months post-challenge.
7. Agreement to refrain from blood donation during the course of the study and for 1 year after the end of their involvement in the study.
8. Willing to take a curative antimalarial regimen following challenge.
9. Willing to be admitted in the Hospital for Tropical Diseases for clinical monitoring until antimalarial treatment (chloroquine) is completed and their symptoms are settling.
10. Willing to reside in Bangkok for the duration of the clinical part of the study, until all antimalarial treatment has been completed.
11. Willing to be followed up for 1 year post treatment initiation.
12. Reachable (24/7) by mobile phone during the period between challenge CHMI and completion of all antimalarial treatment.
13. Able to read and write in Thai and able to answer ALL questions on the informed consent questionnaire correctly.
14. Provided written informed consent to participate in the trial.
15. Cardiovascular risk assessment is low (less than 10% in the next 10 years according to the cardiovascular risk assessment from Thai NCD Division, DDC, MoPH (2016)
16. Educational level: has at least an undergraduate degree.

The volunteer MUST NOT enter the study if any of the following apply:

1. History of clinical malaria.
2. Positive malaria PCR OR malaria film OR malaria serology (recent exposure by Multiplex Bead Based Immunoassay)
3. History of severe allergy to mosquito bite
4. G6PD mutation
5. Presence of any medical condition (either physical or psychological) which in the judgment of the investigator would place the participant at undue risk or interfere with the results of the study (e.g. serious underlying cardiac, renal, hepatic or neurological disease; severe malnutrition; congenital defects or febrile condition)
6. Presence of chronic disease or chronically use of medication.
7. Plan to travel outside of Bangkok within the period of challenge until 3 months after.
8. Use of systemic antibiotics with known antimalarial activity in the 30 days before challenge (e.g. trimethoprim-sulfamethoxazole, doxycycline, tetracycline, clindamycin, erythromycin, fluoroquinolones and azithromycin).
9. Use of immunoglobulins or blood products (e.g. blood transfusion) at any time in the year preceding enrolment.
10. Receipt of an investigational product or any vaccine in the 30 days preceding enrolment (D0), or planned receipt during the study period.
11. Prior receipt of an investigational vaccine likely to impact on interpretation of the trial data or the P. vivax parasite as assessed by the Investigator.
12. Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection, asplenia, history of splenectomy, recurrent, severe infections, and chronic infection.
13. Immunosuppressant medication within the past 6 months preceding enrolment (D0) (inhaled and topical steroids are allowed).
14. History of allergic disease or reactions likely to be exacerbated by malaria infection.
15. Female participant who is pregnant and, lactating during the course of the study, or planning pregnancy within 1 year post-challenge.
16. Contraindications to the use of antimalarial treatment (e.g. chloroquine or primaquine or atovaquone / proguanil, DHA piperaquine).
17. Use of medications known to have a potentially clinically significant interaction with antimalarial drug that will be used in this study (chloroquine or primaquine or atovaquone / proguanil, DHA/ piperaquine).
18. Use of medications known to cause prolongation of the QT interval as state in the section of prohibited drugs that may have effect on prolongation of the QT interval.*
19. Known existing positive family history in both 1st AND 2nd degree relatives < 50 years old for cardiac disease.
20. Family history of congenital QT prolongation or sudden death.
21. Any clinical condition known to prolong the QT interval.
22. History of cardiac arrhythmia, including clinically relevant bradycardia.
23. Screening ECG demonstrates a QTc interval ≥ 450 ms
24. Suspected or known or history of alcohol abuse
25. Suspected or known or history of drug abuse.
26. Concurrently participating in another clinical study, at any time during the study period.
27. Finding on safety laboratory values as defined below:

    * Abnormal ALT [>upper normal range]
    * Abnormal serum creatinine [>upper normal range]
    * Clinically significant abnormalities in corrected calcium and magnesium blood levels
    * Haemoglobin < 11 g/dL
    * HbA1C >upper normal range
28. Thalassaemia disease or haemoglobinopathies.
29. Positive hepatitis B surface antigen or seropositive for hepatitis C virus, or HIV, Syphilis, HTLVI/II

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
The minimum number of infected mosquito bites. | Up to 21 days after the individual CHMI
  The minimum number of infected mosquito bites needed to reliably result in a P.vivax infection in all 12 participants at a given bite dose group, as defined by two consecutive positive qPCR results or presence of parasitemia on malaria blood film

SECONDARY OUTCOMES:
Prepatent period across different groups. | Up to 21 days after the individual CHMI
  Measurement of the prepatent period (time from challenge to first qPCR-positive result) in participants across different mosquito bite groups.
Humoral immune responses | Up to one year after antimalarial initiation
  Characterisation of humoral immune responses (antibody titress) to Plasmodium vivax infection, stratified by the number of mosquito bites received.
Humoral immune responses | Up to one year after antimalarial initiation
  Characterisation of humoral immune responses (Cytokine response) to Plasmodium vivax infection, stratified by the number of mosquito bites received.
Cellular immune responses | Up to one year after antimalarial initiation
  Characterisation of cellular immune responses (T-cell profiles) to Plasmodium vivax infection, stratified by the number of mosquito bites received.
Cellular immune responses | Up to one year after antimalarial initiation
  Characterisation of cellular immune responses (Neutrophil) to Plasmodium vivax infection, stratified by the number of mosquito bites received.
Gametocytaemia across different groups | Up to 21 days after the individual CHMI
  Quantification of gametocytaemia measured by quantitative PCR (qPCR) across different groups
AEs stratified by groups | Up to one year after antimalarial initiation
  Incidence, severity, and duration of AEs stratified by number of mosquito bites administered.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Day, MD, Principal Investigator — University of Oxford; Jetsumon Sattabongkot Prachumsri, Ph.D, Principal Investigator — Mahidol University
Locations (1):
- Faculty of Tropical Medicine, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
With participant's consent, suitably anonymised clinical data and results from blood analyses stored in the database may be shared according to the terms defined in the MORU data sharing policy with other researchers to use in the future.
Supporting Information: Study Protocol, SAP
Time Frame: After completion of trial activities and once the study data have already been used for the study purposes, including publication.
URL: https://www.tropmedres.ac/units/moru-bangkok/bioethics-engagement/data-sharing